CLINICAL TRIAL: NCT01116206
Title: A Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Prucalopride (Resolor) Tablets in Participants With Chronic Constipation
Brief Title: An Efficacy and Safety Study of Prucalopride in Participants With Chronic Constipation
Acronym: Resolor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017173; PRUCRC3001 (Other Grant/Funding Number: Johnson & Johnson Pharmaceutical Research and Development, L.L.C)
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Constipation
Keywords: Constipation; Prucalopride; Resolor
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prucalopride (Experimental): prucalopride 2- milligram (mg), orally once daily for 12 weeks
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Matching placebo, orally once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — 2 mg tablet, orally once daily, for 12 weeks
  Other Names: Resolor
  Arms: Prucalopride
Drug: Placebo — 1 tablet, orally once dailyfor 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of prucalopride to placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) in treatment of participants with chronic (very serious, life threatening) constipation (decreased number of or difficulty making bowel [the intestine] movements).

DETAILED DESCRIPTION:
This is a randomized (study drug is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participants receives), placebo-controlled, multi-center (when more than 1 hospital or medical school team work on a medical research study) study with a parallel-group design (a medical research study comparing the response in 2 or more groups of participants receiving different treatments) study of prucalopride. This study consist of 3 phases: a 2 weeks drug-free screening or run in phase, a 12-week treatment phase and follow-up (post-treatment) phase performed 7 days following the last dose of study drug. The total duration of study will be approximately 15 to 20 weeks, including the run-in and post-treatment phases. During the run-in phase, participants will receive laxative (bisacodyl) as a rescue medication throughout the study, if they will not have bowel movement (BM) for 3 or more consecutive days. If participants will not be able to tolerate bisacodyl, an enema may be used in place of the bisacodyl. During the double-blind treatment phase, participants will be randomly assigned in a 1:1 ratio to 1 of 2 treatment groups to receive either 2 milligram (mg) prucalopride or matching placebo prucalopride for 12 weeks, orally once daily. Participants will be primarily assessed for spontaneous complete bowel movements (SCBMs) per week. Participant's safety and quality of life will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic constipation, defined as on average, 2 or fewer spontaneous bowel movements (SBMs) per week and 1 or more of the following for at least a quarter of the time for the last 3 months, while symptom onset was more than 6 months before the screening visit: in more than 25 percent (%) of BMs, participants had very hard (little balls) and/or hard stools, sensation of incomplete evacuation, straining at defecation (making a bowel movement), sensation of ano-rectal obstruction or blockade, and/or need for digital manipulation to facilitate evacuation
* Participants who were considered as constipated (who never had SBMs)
* Participant's constipation is functional
* Participants with the diagnosis of irritable bowel syndrome (bowel disorder in which there is pain and diarrhea or constipation) with constipation and with no other organic diseases can potentially be included depending on the decision of the investigator
* Female participants must be postmenopausal (for at least 1 year) or surgically sterile or practicing a highly effective method of birth control

Exclusion Criteria:

* Secondary to other diseases/conditions (endocrine disorders, metabolic disorders or neurologic disorders or drug-induced or suspected organic disorders of the large bowel, i.e., obstruction, carcinoma (type of cancer), or inflammatory bowel disease)
* - Participants Using or intending to use disallowed medications that may influence the bowel habit during the study
* Participants with severe (very serious, life threatening) and clinically uncontrolled cardiovascular, liver, or lung disease, neurologic or psychiatric disorders (including active alcohol or drug abuse), cancer (abnormal tissue that grows and spreads in the body until it kills) or acquired immune deficiency syndrome (AIDS: illness that results in decreased ability of the body to protect itself from other illnesses; development of the disease or conditions associated with the disease results from Human Immunodeficiency Virus [HIV]), or other gastrointestinal or endocrine disorders
* Participants with impaired renal function, that is, serum creatinine greater than 2 milligram per deciliter (greater than 180 micro mole per liter)
* Participants with clinically significant abnormalities of hematology, urinalysis, or blood chemistry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With an Average of 3 or More Spontaneous Complete Bowel Movements (SCBMs) | Week 1 to 12
  Percentage of responders (responders: participants with an average of 3 or more SCBMs per week) will be assessed during 12-week double-blind treatment phase (total treatment duration). SCBM is defined as a Spontaneous Bowel Movement (SBM) associated with a sense of complete evacuation. SBM is defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository used on either the calendar day of the BM or the calendar day before the BM. The total number of SBMs associated with a feeling of complete evacuation will be summed and divided by 12. Average weekly frequency of SCBMs will be calculated as number of SCBMs in treatment phase multiplied by 7 divided by total number of evaluable days in treatment phase.

SECONDARY OUTCOMES:
Percentage of Participants With an Average of 3 or More SCBMs During the First 4 Weeks | Week 1 to 4
  Percentage of responders (participants with an average of 3 or more SCBMs per week) will be assessed during first 4 weeks of 12-week double-blind treatment phase (total treatment duration). SCBM will be defined as a Spontaneous Bowel Movement (SBM) associated with a sense of complete evacuation. SBM is defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository used on either the calendar day of the BM or the calendar day before the BM. Average weekly frequency of SCBMs will be calculated as number of SCBMs in Week 1 to 4 multiplied by 7 divided by total number of evaluable days in Week 1 to 4.
Percentage of Participants With an Average Increase of 1 or More Bowel Movements (BMs) | Week 1 to 12
  Percentage of participants with an average increase of 1 or more SCBMs per week as compared to the run-in phase (that is screening phase at Week Minus 2) will be assessed. SCBM is defined as SBM that is associated with a sense of complete evacuation. SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Average weekly frequencies will be calculated as number of SCBMs in interval multiplied by 7 divided by total number of evaluable days in interval.
Percentage of Participants With an Average of 3 or More SCBMs During Weeks 5 to 8 and 9 to 12 | Week 5 to Week 8 and Week 9 to Week 12
  Percentage of participants with an average increase of 3 or more SCBMs per week will be assessed. SCBM is defined as SBM that is associated with a sense of complete evacuation. SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Average weekly frequencies will be calculated as number of SCBMs in interval multiplied by 7 and divided by total number of evaluable days in interval.
Average Number of SCBMs | Week 1 to 12
  An increase in the average number of SCBMs per week will be assessed during Weeks 1 to 12. SCBM will be defined as a SBM that is associated with a sense of complete evacuation. SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Average weekly frequencies will be calculated as (number of SCBMs in interval * 7) / number of evaluable days in interval.
Average Number of Spontaneous Bowel Movements (SBMs) | Week 1 to 12
  Average number of SBMs is assessed. SBM is defined as a BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Average weekly frequencies will be calculated as (number of SBMs in interval * 7) / number of evaluable days in interval.
Average Number of all Bowel Movements (BMs) | Week 1 to 12
  Average number of BMs will be assessed.BMs are spontaneous discharge of waste matterfrom the large intestine. Average weekly frequencies will be calculated as (number of BMs in interval * 7) / number of evaluable days in interval.
Time-to-First SCBM and Time-to-First Week With 3 or More SCBMs After the First Dose of the Study Drug | Week 1 to 12
  SCBM is defined as a SBM that is associated with a sense of complete evacuation. SBM is defined as a bowel movement BM that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM. Average weekly frequencies will be calculated as (number of SCBMs in interval * 7) / number of evaluable days in interval.
Average Number of Bisacodyl Tablets | Week 1 to 12
  Average number of bisacodyl tablets taken is determined. Bisacodyl 5, 10, or 15 milligram (mg) is used as rescue medication. Rescue medications are medicines that may be administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Average weekly frequencies will be calculated as (number of bisacodyl tablets in interval * 7) / number of evaluable days in interval.
Percentage of Participants With Zero, Less Than (<) 2 and Greater Than and Equal to (>=) 2 Tablets of Bisacodyl Taken | Week 1 to 12
  Average number of bisacodyl tablets taken will be determined during 12-week double-blind treatment phase. Bisacodyl 5, 10, or 15 milligram (mg) will be used as rescue medication. Rescue medications are medicines that may be administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Average weekly frequencies will be calculated as (number of bisacodyl tablets in interval * 7) / number of evaluable days in interval.
Percentage of BMs With Normal Consistency | Week 1 to 12
  Percentage of BM with normal consistency for each participant will be calculated by dividing number of BMs with normal consistency with total number of BMs in that participant multiplied by 100. Average of percentage of BM with normal consisitency for all participants have been reported. The consistency of each BM will be assessed using the 7-point Bristol Stool Scale: score ranging from 1 to 7,wherein 1=stool is separate hard lumps, like nuts (hard to pass); and 7=watery, no solid pieces, entirely liquid (passed easily). Score 3 and 4 indicates normal consistency.
Percentage of BMs With Less Straining | Week 1 to 12
  Percentage of BM with less straining for each participant will be calculated by dividing number of BMs with less straining with total number of BMs in that participant multiplied by 100. Average of percentage of BM with less straining for all participants will be reported. Degree of straining is measured on a 5-point scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe. Less straining indicates none or mild degree of straining.
Percentage of BMs with a Sensation of Complete Evacuation | Week 1 to 12
  Percentage of BM with a sensation of complete evacuation for each participant will be calculated by dividing number of BMs with a sensation of complete evacuation with total number of BMs in that participant multiplied by 100. Average of percentage of BM with a sensation of complete evacuation for all participants will be reported. Percentage of BMs with a sensation of complete evacuation will be calculated as (number of BMs with a sensation of complete evacuation in interval / [number of SCBMs or BMs with non - missing scores in interval] * 100%).
Participants Global Assessment on Consistency of Stool | Week 2, 4, 8 and 12
  Participants Global Assessment on consistency of stool will be assessed with Types 1-2=constipation,Types 3-4= ideal stools and Types 5-7=further tending towards diarrhea or urgency based on Bristol Stool Scale. Bristol Stool Scale:1=stool is separate hard lumps, like nuts (hard to pass);2=stool is sausage-shaped but lumpy; 3=stool is like a sausage but with cracks on its surface; 4=stool is like a sausage or snake, smooth and soft; 5=stool is soft blobs with clear-cut edges (passed easily);6=fluffy pieces with ragged edges, mushy stool;7=watery, no solid pieces, entirely liquid (passed easily).
Participants Global Assessment on Severity of Constipation | Week 2, Week 4, Week 8 and Week 12
  Participants Global Assessmentof severity of constipation will be assessed using a 5-point scale ranging from 0 to 4: 0=absent (no constipation); 1=mild constipation; 2=moderate constipation; 3=severe constipation; 4=very severe constipation.
Participants Global Assessment on Efficacy of Treatment | Week 2, Week 4, Week 8, and Week 12
  Participants global assessment on efficacy of treatment was assessed using a 5-point scale ranging from 0 to 5: 0=not at all effective; 1=a little bit effective; 2=moderately effective; 3=quite a bit effective; 4=extremely effective.
Investigator's Global Assessment on Efficacy of Treatment | Week 4 and 12
  Investigator's Global Assessment on efficacy of treatment will be assessed using rating on a 5-point scale: 0=not at all effective; 1=a little bit effective; 2=moderately effective; 3=quite a bit effective; 4=extremely effective
Change From Baseline in Patient Assessment of Constipation-Symptom Questionnaire (PAC-SYM) Total Score at Week 2, 4, 8 and 12 | Baseline, Week 2, 4, 8, and 12
  The PAC-SYM is a 12-item participant self-administered instrument that measures the severity of constipation-related symptoms. Items are rated on a 5-point Likert scale, where 0=absent, 1=mild, 2=moderate, 3=severe, and 4=very severe. The PAC-SYM contains 3 subscales: stool symptoms (5 items), abdominal symptoms (4 items) and rectal symptoms (3 items)
Change From Baseline in the PAC-SYM Subscale Scores at Week 2, 4, 8 and 12 | Baseline, Week 2, 4, 8, and 12
  The PAC-SYM is comprised of the following 3 subscales: Stool symptoms (5 items): bowel movements that require straining or squeezing, bowel movements that are too hard, bowel movements that are too small, bowel movements that result in a sensation of incomplete evacuation, the feeling of having to pass a bowel movement but couldn't (false alarm); Abdominal symptoms (4 items):abdominal discomfort, abdominal pain, abdominal cramping, abdominal bloating; Rectal symptoms (3 items): painful bowel movements, rectal burning, bleeding or tearing during or after a bowel movement.
Percentage of Participant's who Rated Study Drug effectiveness | Week 2, Week 4, Week 8 and Week 12
  The percentage of participants who rated the study treatment with efficacy score of 3=quite a bit to 4=extremely effective on global evaluation of efficacy of treatment was determined.
Percentage of Participants With PAC SYM Score | Weeks 2, 4, 8, and 12
  Percentage of participants with an improvement of greater than or equal to 1 point on the PAC SYM score will be determined. The PAC-SYM is a 12-item participant self-administered instrument that measures the severity of constipation-related symptoms. Items are rated on a 5-point Likert scale, where 0=absent, 1=mild, 2=moderate, 3=severe, and 4=very severe. The PAC-SYM contains 3 subscales: stool symptoms (5 items), abdominal symptoms (4 items) and rectal symptoms (3 items).

OTHER OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Week 13
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 7 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Number of Participants With Clinically Significant Laboratory Values | Baseline up to Week 12
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.
Number of Participants With Clinically Significant Vital Signs Abnormalities | Baseline up to Week 12
  Number of participants with potentially clinically important (PCI) vital signs is reported during therapy and at post therapy. Criteria for PCI change in vital signs: pulse rate value is defined as : low (decrease from baseline of >= 15 to a value =< 50) and high (increase from baseline of >= 15 to a value >=120), systolic blood pressure (SBP) is defined as: low (decrease from baseline of >= 20 to a value =< 90) and high (increase from baseline of >= 20 to a value >=180), diastolic blood pressure (DBP) is defined as: low (decrease from baseline of >=15 to a value =<50) and high (increase from baseline of >= 15 to a value >=105).
Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities | Baseline up to Week 12
  Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum increase from baseline of 30 to less than (<) 60 msec(borderline) and greater than or equal to (>=) 60 msec (prolonged) were summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (27):
- Australia (8):
  - Adelaide
  - Box Hill
  - Kingswood
  - Kogarah
  - Newcastle
  - Parkville
  - Prahran
  - Sydney
- China (10):
  - Beijing
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Hefei
  - Jinan
  - Nanjing
  - Shanghai
  - Wuhan
  - Xi'an
- South Korea (6):
  - Busan
  - Daegu
  - Deajun
  - Gwangju
  - Iksan
  - Seoul
- Taipei, Taiwan
- Thailand (2):
  - Bamgkok
  - Bangkok

REFERENCES:
- [Derived] Lembo A, Staller K, Boules M, Feuerstadt P, Spalding W, Gabriel A, Youssef A, Xie Y, Terreri B, Cash BD. Efficacy and safety of prucalopride in patients with chronic idiopathic constipation stratified by age, body mass index, and renal function: a post hoc analysis of phase III and IV, randomized, placebo-controlled clinical studies. Therap Adv Gastroenterol. 2024 Dec 10;17:17562848241299731. doi: 10.1177/17562848241299731. eCollection 2024. PMID 39664231
- [Derived] Staller K, Hinson J, Kerstens R, Spalding W, Lembo A. Efficacy of Prucalopride for Chronic Idiopathic Constipation: An Analysis of Participants With Moderate to Very Severe Abdominal Bloating. Am J Gastroenterol. 2022 Jan 1;117(1):184-188. doi: 10.14309/ajg.0000000000001521. PMID 34585675
- See also: A Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Prucalopride (Resolor) Tablets in Subjects with Chronic Constipation — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=852&filename=CR017173_CSR.pdf